CLINICAL TRIAL: NCT02182414
Title: Relative Bioavailability of BI 207127 Trial Formulation II Prototypes Versus BI 207127 Trial Formulation I Administered Orally as Tablet in Single Doses of 800 mg to Healthy Volunteers, and Evaluation of the Effect of Food on the Bioavailability of a Selected Prototype (an Open-label, Two-stage, Within Parts Randomised Six-way and Two-way Crossover Phase I Study)
Brief Title: Relative Bioavailability of BI 207127 Trial Formulation II Prototypes Versus BI 207127 Trial Formulation I in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1241.9
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (8):
- BI 207127 NA (TF-I) (Active Comparator): trial part 1: 800 mg BI 207127 NA Trial formulation I (TF-I)
  Interventions: Drug: BI 207127 NA (TF-I)
- BI 207127 NA (TF-II) (Experimental): trial part 1: 800 mg BI 207127 NA Trial formulation II (TF-II)
  Interventions: Drug: BI 207127 NA (TF-II)
- BI 207127 NA delayed release (Experimental): trial part 1: 800 mg BI 207127 NA TF-II, delayed release
  Interventions: Drug: BI 207127 NA delayed release
- BI 207127 NA extended release (10% HPMC) (Experimental): trial part 1: 800 mg BI 207127 NA TF-II, extended release (10% Hydroxypropyl methyl cellulose (HPMC))
  Interventions: Drug: BI 207127 NA extended release (10% HPMC)
- BI 207127 NA extended release (15% PEO) (Experimental): trial part 1: 800 mg BI 207127 NA TF-II, extended release (15% Polyethylene oxide (PEO))
  Interventions: Drug: BI 207127 NA extended release (15% PEO)
- BI 207127 NA extended release (20% HPMC) (Experimental): trial part 1: 800 mg BI 207127 NA TF-II, extended release (20% HPMC)
  Interventions: Drug: BI 207127 NA extended release (20% HPMC)
- BI 207127 (TF-II), fed (Experimental): trial part 2
  Interventions: Drug: BI 207127 NA (TF-II); Drug: BI 207127 NA delayed release; Drug: BI 207127 NA extended release (10% HPMC); Drug: BI 207127 NA extended release (15% PEO); Drug: BI 207127 NA extended release (20% HPMC)
- BI 207127 (TF-II), fasted (Experimental): trial part 2
  Interventions: Drug: BI 207127 NA (TF-II); Drug: BI 207127 NA delayed release; Drug: BI 207127 NA extended release (10% HPMC); Drug: BI 207127 NA extended release (15% PEO); Drug: BI 207127 NA extended release (20% HPMC)

INTERVENTIONS:
Drug: BI 207127 NA (TF-I) — 200 mg tablet
  Arms: BI 207127 NA (TF-I)
Drug: BI 207127 NA (TF-II) — 400 mg tablet
  Arms: BI 207127 (TF-II), fasted; BI 207127 (TF-II), fed; BI 207127 NA (TF-II)
Drug: BI 207127 NA delayed release — 400 mg tablet
  Arms: BI 207127 (TF-II), fasted; BI 207127 (TF-II), fed; BI 207127 NA delayed release
Drug: BI 207127 NA extended release (10% HPMC) — 400 mg tablet
  Arms: BI 207127 (TF-II), fasted; BI 207127 (TF-II), fed; BI 207127 NA extended release (10% HPMC)
Drug: BI 207127 NA extended release (15% PEO) — 400 mg tablet
  Arms: BI 207127 (TF-II), fasted; BI 207127 (TF-II), fed; BI 207127 NA extended release (15% PEO)
Drug: BI 207127 NA extended release (20% HPMC) — 400 mg tablet
  Arms: BI 207127 (TF-II), fasted; BI 207127 (TF-II), fed; BI 207127 NA extended release (20% HPMC)

SUMMARY:
Study to investigate the relative bioavailability of 5 new 400 mg tablet formulations (trial formulation II prototypes) of BI 207127 compared to the current 200 mg BI 207127 tablet formulation (trial formulation I) in healthy male volunteers with the aim to identify the best formulation for further drug development (formulation finding part / trial part 1) and to investigate the effect of food on the relative bioavailability of the most promising one of these trial formulation II prototypes (food-effect part / trial part 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to a complete medical history, including a physical examination,vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age 18 to 50 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month prior to administration of the trial drug or during the trial
* Use of any drugs (including herbal preparations, vitamins and nutrient supplements) within 14 days prior to first administration of the trial drug or during the trial
* Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to first administration of the trial drug or during the trial)
* Excessive physical activities (within one week prior to first administration of the trial drug of the trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 MS)
* A history of additional risk factors for Torsade de Points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* History of photosensitivity or recurrent rash

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for BI 207127 | up to 48 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) for BI 207127 | up to 48 hours after drug administration

SECONDARY OUTCOMES:
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval from t1 to t2) | up to 24 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
λz (terminal rate constant in plasma) | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after p.o. administration) | up to 48 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 hours after drug administration
The fluctuation parameter Cmax/C12 for the ER (Extended release) formulations only | up to 48 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 24 hours after drug administration in the food-effect part
fet1-t2 (fraction of analyte eliminated in urine compared to oral dose administered from time point t1 to time point t2) | up to 24 hours after drug administration in the food-effect part
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 24 hours after drug administration in the food-effect part
RCmax,Met (the ratio of Cmax of the metabolite, CD 6168 to Cmax of the parent compound, BI207127) | up to 48 hours after drug administration
RAUC0-∞,Met (the ratio of AUC0-∞ of the metabolite, CD 6168 to AUC0-∞ of the parent compound, BI207127) | up to 48 hours after drug administration
AUC0-∞ for CD 6168 | up to 48 hours after drug administration
Cmax for CD 6168 | up to 48 hours after drug administration
Measurement of protein binding in human plasma for BI 207127 | up to 48 hours after drug administration in the food-effect part
Number of patients with adverse events | up to 9 weeks
Assessment of tolerability on a 4-point scale | 48 h after each drug administration